CLINICAL TRIAL: NCT07236203
Title: Predictive Factors for the Efficacy of CD19 CAR-T Therapy in Relapsed/Refractory Large B-Cell Lymphoma: A Clinical Study
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Rong Tao, Professor, Fudan University
Other Study IDs: CD19 CAR-T
Record Dates: First submitted 2025-05-25; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Large B-Cell Lymphoma
Keywords: CD19 CAR-T; Recurrent/Refractory Large B-Cell Lymphoma; Predictive factors for therapeutic efficacy
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: CAR-T
  Interventions: Drug: CAR-T

INTERVENTIONS:
Drug: CAR-T — CD19 CAR-T

SUMMARY:
This is a single-center real-world study aiming to explore predictive factors for the efficacy of CAR-T therapy in patients with relapsed/refractory large B-cell lymphoma (R/R LBCL).

DETAILED DESCRIPTION:
This single-center, prospective, single-arm phase II observational study aims to investigate multidimensional correlations between clinical baseline characteristics, tumor biological profiles, dynamic changes in CAR-T cell subsets, immune microenvironment features, and therapeutic outcomes in patients with relapsed/refractory diffuse large B-cell lymphoma (LBCL). The study will enroll 80 participants who will receive a standardized 90-day CAR-T therapy regimen. Post-intervention management will be stratified based on the results of treatment efficacy and transplant evaluation: patients failing to achieve complete remission (CR) or exhibiting progressive disease (PD) during therapy may receive investigator-determined salvage therapies, while responders will transition to long-term follow-up. The primary endpoint is to explore predictors of CAR-T efficacy through multivariate analysis of patients' clinical baseline characteristics, tumor characteristics, CAR-T cell subsets and their dynamic changes, and immune microenvironment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis confirmed as large B-cell lymphoma
2. Patients with relapsed or refractory large B-cell lymphoma (R/R DLBCL) after receiving second-line or above systemic treatment
3. Intend to use CAR-T products approved by NMPA for the treatment of R/R LBCL.
4. Understand and voluntarily sign a written informed consent form. For patients without full civil capacity, their guardians must be informed and sign the corresponding informed consent form and note the date, as for the patient himself, informed consent may be obtained based on the specific circumstances.

Exclusion Criteria:

1. Poor patient compliance
2. During pregnancy or lactation
3. After judgment by the researcher, the patient has other unsuitable conditions for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators identified patients with Relapsed/refractory large B-cell lymphoma who could be used and who were willing to receive CAR-T
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
explore predictors of CAR-T efficacy | Baseline; 30 days post-infusion, 90 days post-infusion
  explore predictors of CAR-T efficacy through multivariate analysis of patients' clinical baseline characteristics, tumor characteristics, CAR-T cell subsets and their dynamic changes, and immune microenvironment.

CONTACTS AND LOCATIONS:
Overall Officials: Chuan xu Liu, M.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No